CLINICAL TRIAL: NCT00899392
Title: Improving Informed Consent and Assent in Pediatric Endoscopy
Brief Title: Improving Informed Consent in Pediatric Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Midwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008-6-6053
Record Dates: First submitted 2009-05-08; First posted 2009-05-12 (Estimated); Results first posted 2013-07-30 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Informed Consent; Procedural State Anxiety; Subject's Satisfaction
Keywords: consent; Anxiety; Satisfaction; Efficiency; Questions; Attainment of Informed Consent (Consent-20); Procedural State Anxiety (STAI); Subject Satisfaction (mGHAA-9); Duration in Endoscopy Suite; Number of questions asked
MeSH Terms: conditions — Anxiety Disorders; Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electronic Assisted Consent (Experimental): Standard procedural consent performed by pediatric gastroenterologist plus assistance from computerized emmi module.
  Interventions: Other: Emmi Pediatric Upper Endoscopy Patient Education Module
- Control Consent (No Intervention): Standard procedural consent as performed by pediatric gastroenterologists

INTERVENTIONS:
Other: Emmi Pediatric Upper Endoscopy Patient Education Module — Emmi Pediatric Upper Endoscopy Patient Education Module as designed by EMMI SOLUTIONS, LLC
  Other Names: Pediatric Upper Endoscopy Patient Education Module; Patient Education Module; Upper Endoscopy Patient Education Module; Endoscopy Patient Education Module
  Arms: Electronic Assisted Consent

SUMMARY:
Informed consent/assent in pediatric medicine is an accepted and important practice that has been rarely studied, tested for quality, or optimized for patient satisfaction. In the pursuit of enhancing and studying pediatric care, the investigators propose, as pediatric gastroenterologists, assessing the current state of parental and adolescent consent/assent in upper gastrointestinal endoscopy and offering a computer based education program to improve it. The investigators will look at outcomes that include anxiety, satisfaction, attainment of informed consent, and patient flow efficiency in a GI endoscopy suite.

DETAILED DESCRIPTION:
Two hundred first-time upper endoscopy patients from The Children's Hospital of Philadelphia will be prospectively selected for participation in the study. One hundred subjects will then be randomized to participate in either the standard consent arm or the electronic assisted informed consent (EAIC) arm. The electronic assisted informed consent web module is a professionally designed program by Emmi Solutions, LLC. Adolescents, if present and greater than 13 years of age, will undergo the program apart from their parent as a separate subgroup not included in the 100 randomized subjects. At time of endoscopy scheduling, the scheduler will ask the subjects if they would like to participate in the study. If interest is expressed the study coordinator or PI will contact the subject to explain the study and inform them of the study parameters. At time of phone contact, consent or assent via a verbal method will be performed. Once verbal consent is given by the subject or verbal assent by the adolescent subject they will follow the protocol. No incentives will be given to the subjects. Institutional Review Board (IRB) approval will be obtained.

Between 24 and 48 hours prior to endoscopy, the participant will have the option to access the web-based module outside the hospital or through a hospital-based kiosk. The web address used is http://www.pedsgiconsent.com. Just prior to starting the module, a five-minute electronic pre-intervention test will be given and its results recorded in an electronic database. This will gather demographic and pre-intervention state anxiety without personal identifying information. After the survey is complete, the educational module will be accessed. Upon completion, the subjects will print a confirmatory document of completion and a list of questions to hand to their physician at time of endoscopy. Hand written questions will also be permitted. Non-EAIC participants will perform a non-educational web program not related to gastroenterology and also have their endoscopy questions printed to give to their physician. The questions and confirmation sheet will also be presented to their physician at time of procedure. Participants will also have space to write further questions by hand on the form. The questions collected will be used to assess number and complexity of questions asked as influenced by the education program. The web module will record time duration taken for the program. After completing the program, the participants will report to the GI suite as previously scheduled. The procedure will occur without either the practitioner or nursing staff knowing in which arm of the study the participants are enrolled. After the questions are answered and formal GI endoscopy procedural consent is obtained, the question sheet will be deposited in a lock box in the endoscopy suite for review at a later time. Total time spent in the endoscopy suite will be recorded. Prior to the patient's endoscopy, but after formal consent is obtained, the participant will then take a ten minute electronic post-test to ascertain satisfaction (mGHAA-modified-Group Health Association of America Survey-9), change in state anxiety [s-STAI-(Spielberger-State Trait Anxiety Inventory (state section)], and change in understanding of consent parameters achieved. Satisfaction will be measured using the validated modified Group Health Association of America-9 Survey (mGHAA-9). It is a well-validated instrument used to measure patient satisfaction in adult endoscopy. Probing questions to evaluate the attainment of consent will be based on a modified survey taken from Woodrow's study titled, "How Thorough is the Process of Informed Consent Prior to Outpatient Gastroscopy?"(Consent-20)

ELIGIBILITY:
Inclusion Criteria:

* Parent of child undergoing 1st, elective, outpatient, sedated, upper endoscopy (EGD)
* Subject gives consent to participate
* Child of parent does not have a planned endoscopy intervention.

Exclusion Criteria:

* Does not speak or understand English
* Does not give consent to participate
* Does not complete consent instrument at a minimum during study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2008-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Petar Mamula, M.D., Principal Investigator — Children's Hospital of Philadelphia; Joel Friedlander, D.O., M.Be., Principal Investigator — Children's Hospital of Phildelphia; Greg Loeben, Ph.D., Study Chair — Midwestern University
Locations (1):
- Chidren's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Woodrow SR, Jenkins AP. How thorough is the process of informed consent prior to outpatient gastroscopy? A study of practice in a United Kingdom District Hospital. Digestion. 2006;73(2-3):189-97. doi: 10.1159/000094528. Epub 2006 Jul 11. PMID 16837805
- [Background] Gros DF, Antony MM, Simms LJ, McCabe RE. Psychometric properties of the State-Trait Inventory for Cognitive and Somatic Anxiety (STICSA): comparison to the State-Trait Anxiety Inventory (STAI). Psychol Assess. 2007 Dec;19(4):369-81. doi: 10.1037/1040-3590.19.4.369. PMID 18085930
- [Background] Yacavone RF, Locke GR 3rd, Gostout CJ, Rockwood TH, Thieling S, Zinsmeister AR. Factors influencing patient satisfaction with GI endoscopy. Gastrointest Endosc. 2001 Jun;53(7):703-10. doi: 10.1067/mge.2001.115337. PMID 11375575
- [Background] Standards of Practice Committee; Zuckerman MJ, Shen B, Harrison ME 3rd, Baron TH, Adler DG, Davila RE, Gan SI, Lichtenstein DR, Qureshi WA, Rajan E, Fanelli RD, Van Guilder T. Informed consent for GI endoscopy. Gastrointest Endosc. 2007 Aug;66(2):213-8. doi: 10.1016/j.gie.2007.02.029. No abstract available. PMID 17643691
- [Derived] Friedlander JA, Loeben GS, Finnegan PK, Puma AE, Zhang X, de Zoeten EF, Piccoli DA, Mamula P. A novel method to enhance informed consent: a prospective and randomised trial of form-based versus electronic assisted informed consent in paediatric endoscopy. J Med Ethics. 2011 Apr;37(4):194-200. doi: 10.1136/jme.2010.037622. Epub 2011 Jan 18. PMID 21245476
- See also: The Study Web Site — http://www.pedsgiconsent.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 2008 and March 2009, parents of 220 children scheduled for clinically indicated upper endoscopy were prospectively and consecutively contacted. 190 subjects verbally consented to be in the study and 148 subsequently participated. 6 were withdrawn from data secondary to entering disqualifying demographic response (not in data set)
Pre-assignment Details: 30 subjects did not participate because they did not consent to participate. These were not enrolled in the study.
Groups:
- Electronic Assisted Consent (EAC): Standard form-based procedural consent performed by pediatric gastroenterologist plus assistance from computerized Emmi module.
- Control Consent (FBC): Form-based informed consent as performed by pediatric gastroenterologists
Period: Overall Study
Arm/Group | Electronic Assisted Consent (EAC) | Control Consent (FBC)
Started | 68 | 74
Completed | 47 (Subjects:PerVariableStudied Consent:47-EAC 50-FBC Anxiety:60-EAC 3-FBC Satisfaction:63-EAC 67-FBC) | 50 (Subjects:PerVariableStudied Consent:47-EAC 50-FBC Anxiety:60-EAC 3-FBC Satisfaction:63-EAC 67-FBC)
Not Completed | 21 | 24
Not completed — Subject didn't finish/partial pilot data | 21 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Electronic Assisted Consent (EAC) | Control Consent (FBC) | Total
Number analyzed (Participants) | 68 | 74 | 142
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 68 | 74 | 142
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — EAC population are subjects that used web based education module
  Participants
    Female | 50 | 60 | 110
    Male | 18 | 14 | 32

OUTCOME MEASURES:

1. Primary Outcome: Attainment of Informed Consent as Measured by Consent Instrument (Consent-20)
Description: Units on a scale (score) as Measured by Consent 20 Instrument.
  20 questions administered on a laptop computer and answered in private. Questions 1-5: qualitative questions about recalling procedure, risks, benefits, etc. (correct or incorrectly scored 0 or 2 points), Questions 6-20: yes or no responses, measuring delivery, voluntariness, and understanding. Each scored 0 or 2 points.
  Measures theoretical attainment of a minimum standard of informed consent. Worse value: Zero Best Value: 40
Time Frame: Every 1-2 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Electronic Assisted Consent (EAC) | Control Consent (FBC)
Number analyzed (Participants) | 47 | 50
Units on a scale | 37.36 (2.7) | 33.2 (5.2)
Statistical Analysis 1: Comparison: Electronic Assisted Consent (EAC) vs Control Consent (FBC); Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Student's t test

2. Secondary Outcome: Subject (Parental) Satisfaction as Measured by Modified Group Health Association of America-9 Survey (mGHAA-9)
Description: Worse Value: 5 Best Value 45 Measures satisfaction on a scale per the mGHAA-9. 9 questions administered on a laptop in private.
Time Frame: Every 1-2 months
Population: (Consent Group + some pilot participants to increase power of analysis)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Electronic Assisted Consent (EAC) | Control Consent (FBC)
Number analyzed (Participants) | 63 | 67
Units on a scale | 41.79 (3.6) | 41.46 (3.4)
Statistical Analysis 1: Comparison: Electronic Assisted Consent (EAC) vs Control Consent (FBC); Mann Whitney Test-non parametric; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Subject (Parental) State Anxiety as Measured by the Spielberger-State Trait Anxiety Inventory (s-STAI) (State Section)
Description: s-STAI as a series of question administered by laptop computer in private. 20 questions answered on Likert 4 point scale that varies based on question type. Max score 80.
Time Frame: 12-18 hours (Night before Endoscopy to Day of Endoscopy)
Population: Matched pairs (pre consent and post consent), Pilot data included to increase power analysis
Measure: Mean (Standard Deviation); unit: Units on a Scale (STAI Score)
Arm/Group | Electronic Assisted Consent (EAC) | Control Consent (FBC)
Number analyzed (Participants) | 60 | 63
Units on a Scale (STAI Score)
  Day Before Procedure | 42.17 (14.32) | 37.17 (12.56)
  Moments after consent | 38.77 (12.79) | 33.76 (8.94)
Statistical Analysis 1: Comparison: Electronic Assisted Consent (EAC) vs Control Consent (FBC); Test type: Superiority or Other; p > 0.05, t-test, 2 sided; paired

4. Secondary Outcome: Questions Asked by Subjects (Parents)
Description: Number of questions written down by family and asked of clinician. Question sheet given to nurse in endoscopy suite and deposited in a box.
Time Frame: Questions written by parents during the end of consent process (48-72 hours)
Measure: Mean (Full Range); unit: Questions
Arm/Group | Electronic Assisted Consent (EAC) | Control Consent (FBC)
Number analyzed (Participants) | 60 | 63
Questions | 2.03 [0 to 14] | 3.06 [0 to 9]
Statistical Analysis 1: Comparison: Electronic Assisted Consent (EAC) vs Control Consent (FBC); Test type: Superiority or Other; p = 0.0053, t-test, 2 sided

5. Secondary Outcome: GI Suite Flow Efficiency Measured in 15 Minute Increments
Time Frame: At completion of study
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Electronic Assisted Consent (EAC) | Control Consent (FBC)
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/74
Other Adverse Events (participants affected / at risk) | 0/68 | 0/74

LIMITATIONS AND CAVEATS:
Subjects of study did not all complete secondary outcome measures hence some pilot data was included in 2ndary outcome analysis, New instrument used attempting to validate. Largely female, educated cohort. >60% college educated in both groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No